CLINICAL TRIAL: NCT05186623
Title: Establishment of Prediction Model of Biologics and Small Molecular Agent for Patients With Ulcerative Colitis Using Longitudinal Data
Brief Title: Prediction Model for Response to Biologics and Small Molecular Agent for UC
Status: Recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Byong Duk Ye, Professor, Asan Medical Center
Other Study IDs: 2021-1718
Record Dates: First submitted 2021-12-22; First posted 2022-01-11 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Ulcerative Colitis
Keywords: Response, Vedolizumab, Ustekinumab, Tofacitinib, Multiomics
MeSH Terms: conditions — Colitis, Ulcerative | interventions — vedolizumab; Ustekinumab; tofacitinib

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Genomic DNA, serum, feces, colon tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Patients with confirmed ulcerative colitis: Patients with confirmed ulcerative colitis, who are going to receive vedolizumab therapy (n=100: development cohort n=70 and validation cohort n=30), ustekinumab therapy (n=100: development cohort n=70 and validation cohort n=30), or tofacitinib therapy (n=100: development cohort n=70 and validation cohort n=30), will be enrolled.
  Interventions: Drug: Vedolizumab, Ustekinumab, or Tofacitinib

INTERVENTIONS:
Drug: Vedolizumab, Ustekinumab, or Tofacitinib — Drug administration and prospective follow-up for evaluating response

SUMMARY:
This prospective observational study is going to develop and validate a prediction model of response to biologic agents and small molecular agents for Korean patients with ulcerative colitis.

DETAILED DESCRIPTION:
In this prospective observational study, patients with confirmed ulcerative colitis, who are going to receive vedolizumab, ustekinumab, or tofacitinib will be enrolled after an informed consent. In the screening period, inclusion/exclusion criteria will be checked and if eligible and consented, demographic data, medical history, disease characteristics and disease activity data will be collected. Before drug administration (week 0), baseline lower GI endoscopy will be performed and colon tissues will be collected. Blood sample and fecal sample will also be collected. After induction therapy with each drug, clinical and endoscopic response will be evaluated at week 14 to week 16 and patients will be classified into responders non-responders. Combing clinical data, blood laboratory data, fecal inflammatory biomarker, genetic data, and colonic transcriptomic data, a prediction model for response to induction therapy will be developed and it will be validated in another patient group. Similarly, based on evaluation at week 52, a prediction model for maintenance response will also be developed and validated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established diagnosis of ulcerative colitis based on clinical symptoms, endoscopic features and histopathologic features
* Patients who are going to receive vedolizumab, ustekinumab, or tofacitinib treatment

Exclusion Criteria:

* Not Korean ethnicity by family history
* Inflammatory Bowel Disease Unclassified
* Patients who already received colectomy due to ulcerative colitis

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with an established diagnosis of ulcerative colitis and who are going to receive vedolizumab, ustekinumab, or tofacitinib will be enrolled in this study.
  Patients who give a voluntary informed consent will be eligible.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Response to induction therapy | Week 14 to Week 16
  A decrease from baseline in the total Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1, together with Mayo endoscopic subscore of 0 to 1

SECONDARY OUTCOMES:
Remission to induction therapy | Week 14 to Week 16
  Full Mayo score 0 to 2 + Any component of full Mayo score of 1 or less + Mayo endoscopic subscore of 0 to 1
Complete Mayo endoscopic subscore remission to induction therapy | Week 14 to Week 16
  Mayo endoscopic subscore of 0
Ulcerative colitis endoscopic index of severity remission to induction therapy | Week 14 to Week 16
  Ulcerative colitis endoscopic index of 0 to 1
Response to maintenance therapy | Week 52
  A decrease from baseline in the total Mayo score of at least 3 points and at least 30 percent, with an accompanying decrease in the subscore for rectal bleeding of at least 1 point or an absolute subscore for rectal bleeding of 0 or 1, together with Mayo endoscopic subscore of 0 to 1
Remission to maintenance therapy | Week 52
  Full Mayo score 0 to 2 + Any component of full Mayo score of 1 or less + Mayo endoscopic subscore of 0 to 1
Complete Mayo endoscopic subscore remission to maintenance therapy | Week 52
  Mayo endoscopic subscore of 0
Ulcerative colitis endoscopic index of severity remission to maintenance therapy | Week 52
  Ulcerative colitis endoscopic index of 0 to 1

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xavier RJ, Podolsky DK. Unravelling the pathogenesis of inflammatory bowel disease. Nature. 2007 Jul 26;448(7152):427-34. doi: 10.1038/nature06005. PMID 17653185
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Park SH, Kim YJ, Rhee KH, Kim YH, Hong SN, Kim KH, Seo SI, Cha JM, Park SY, Jeong SK, Lee JH, Park H, Kim JS, Im JP, Yoon H, Kim SH, Jang J, Kim JH, Suh SO, Kim YK, Ye BD, Yang SK; Songpa-Kangdong Inflammatory Bowel Disease [SK-IBD] Study Group. A 30-year Trend Analysis in the Epidemiology of Inflammatory Bowel Disease in the Songpa-Kangdong District of Seoul, Korea in 1986-2015. J Crohns Colitis. 2019 Oct 28;13(11):1410-1417. doi: 10.1093/ecco-jcc/jjz081. PMID 30989166
- [Background] Lee JC, Lyons PA, McKinney EF, Sowerby JM, Carr EJ, Bredin F, Rickman HM, Ratlamwala H, Hatton A, Rayner TF, Parkes M, Smith KG. Gene expression profiling of CD8+ T cells predicts prognosis in patients with Crohn disease and ulcerative colitis. J Clin Invest. 2011 Oct;121(10):4170-9. doi: 10.1172/JCI59255. Epub 2011 Sep 26. PMID 21946256
- [Background] Biasci D, Lee JC, Noor NM, Pombal DR, Hou M, Lewis N, Ahmad T, Hart A, Parkes M, McKinney EF, Lyons PA, Smith KGC. A blood-based prognostic biomarker in IBD. Gut. 2019 Aug;68(8):1386-1395. doi: 10.1136/gutjnl-2019-318343. Epub 2019 Apr 27. PMID 31030191
- [Background] Sandborn WJ. Current directions in IBD therapy: what goals are feasible with biological modifiers? Gastroenterology. 2008 Nov;135(5):1442-7. doi: 10.1053/j.gastro.2008.09.053. Epub 2008 Oct 9. No abstract available. PMID 18848556
- [Background] Rutgeerts P, Sandborn WJ, Feagan BG, Reinisch W, Olson A, Johanns J, Travers S, Rachmilewitz D, Hanauer SB, Lichtenstein GR, de Villiers WJ, Present D, Sands BE, Colombel JF. Infliximab for induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2005 Dec 8;353(23):2462-76. doi: 10.1056/NEJMoa050516. PMID 16339095
- [Background] Feagan BG, Rutgeerts P, Sands BE, Hanauer S, Colombel JF, Sandborn WJ, Van Assche G, Axler J, Kim HJ, Danese S, Fox I, Milch C, Sankoh S, Wyant T, Xu J, Parikh A; GEMINI 1 Study Group. Vedolizumab as induction and maintenance therapy for ulcerative colitis. N Engl J Med. 2013 Aug 22;369(8):699-710. doi: 10.1056/NEJMoa1215734. PMID 23964932
- [Background] Sands BE, Sandborn WJ, Panaccione R, O'Brien CD, Zhang H, Johanns J, Adedokun OJ, Li K, Peyrin-Biroulet L, Van Assche G, Danese S, Targan S, Abreu MT, Hisamatsu T, Szapary P, Marano C; UNIFI Study Group. Ustekinumab as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2019 Sep 26;381(13):1201-1214. doi: 10.1056/NEJMoa1900750. PMID 31553833
- [Background] Sandborn WJ, Su C, Sands BE, D'Haens GR, Vermeire S, Schreiber S, Danese S, Feagan BG, Reinisch W, Niezychowski W, Friedman G, Lawendy N, Yu D, Woodworth D, Mukherjee A, Zhang H, Healey P, Panes J; OCTAVE Induction 1, OCTAVE Induction 2, and OCTAVE Sustain Investigators. Tofacitinib as Induction and Maintenance Therapy for Ulcerative Colitis. N Engl J Med. 2017 May 4;376(18):1723-1736. doi: 10.1056/NEJMoa1606910. PMID 28467869
- [Background] Sands BE, Peyrin-Biroulet L, Loftus EV Jr, Danese S, Colombel JF, Toruner M, Jonaitis L, Abhyankar B, Chen J, Rogers R, Lirio RA, Bornstein JD, Schreiber S; VARSITY Study Group. Vedolizumab versus Adalimumab for Moderate-to-Severe Ulcerative Colitis. N Engl J Med. 2019 Sep 26;381(13):1215-1226. doi: 10.1056/NEJMoa1905725. PMID 31553834
- [Background] Barre A, Colombel JF, Ungaro R. Review article: predictors of response to vedolizumab and ustekinumab in inflammatory bowel disease. Aliment Pharmacol Ther. 2018 Apr;47(7):896-905. doi: 10.1111/apt.14550. Epub 2018 Feb 12. PMID 29430672
- [Background] Dulai PS, Boland BS, Singh S, Chaudrey K, Koliani-Pace JL, Kochhar G, Parikh MP, Shmidt E, Hartke J, Chilukuri P, Meserve J, Whitehead D, Hirten R, Winters AC, Katta LG, Peerani F, Narula N, Sultan K, Swaminath A, Bohm M, Lukin D, Hudesman D, Chang JT, Rivera-Nieves J, Jairath V, Zou GY, Feagan BG, Shen B, Siegel CA, Loftus EV Jr, Kane S, Sands BE, Colombel JF, Sandborn WJ, Lasch K, Cao C. Development and Validation of a Scoring System to Predict Outcomes of Vedolizumab Treatment in Patients With Crohn's Disease. Gastroenterology. 2018 Sep;155(3):687-695.e10. doi: 10.1053/j.gastro.2018.05.039. Epub 2018 May 30. PMID 29857091
- [Background] Ungar B, Kopylov U, Yavzori M, Fudim E, Picard O, Lahat A, Coscas D, Waterman M, Haj-Natour O, Orbach-Zingboim N, Mao R, Chen M, Chowers Y, Eliakim R, Ben-Horin S. Association of Vedolizumab Level, Anti-Drug Antibodies, and alpha4beta7 Occupancy With Response in Patients With Inflammatory Bowel Diseases. Clin Gastroenterol Hepatol. 2018 May;16(5):697-705.e7. doi: 10.1016/j.cgh.2017.11.050. Epub 2017 Dec 7. PMID 29223444
- [Background] Zeissig S, Rosati E, Dowds CM, Aden K, Bethge J, Schulte B, Pan WH, Mishra N, Zuhayra M, Marx M, Paulsen M, Strigli A, Conrad C, Schuldt D, Sinha A, Ebsen H, Kornell SC, Nikolaus S, Arlt A, Kabelitz D, Ellrichmann M, Lutzen U, Rosenstiel PC, Franke A, Schreiber S. Vedolizumab is associated with changes in innate rather than adaptive immunity in patients with inflammatory bowel disease. Gut. 2019 Jan;68(1):25-39. doi: 10.1136/gutjnl-2018-316023. Epub 2018 May 5. PMID 29730603
- [Background] Uzzan M, Tokuyama M, Rosenstein AK, Tomescu C, SahBandar IN, Ko HM, Leyre L, Chokola A, Kaplan-Lewis E, Rodriguez G, Seki A, Corley MJ, Aberg J, La Porte A, Park EY, Ueno H, Oikonomou I, Doron I, Iliev ID, Chen BK, Lui J, Schacker TW, Furtado GC, Lira SA, Colombel JF, Horowitz A, Lim JK, Chomont N, Rahman AH, Montaner LJ, Ndhlovu LC, Mehandru S. Anti-alpha4beta7 therapy targets lymphoid aggregates in the gastrointestinal tract of HIV-1-infected individuals. Sci Transl Med. 2018 Oct 3;10(461):eaau4711. doi: 10.1126/scitranslmed.aau4711. PMID 30282696
- [Background] Schleier L, Wiendl M, Heidbreder K, Binder MT, Atreya R, Rath T, Becker E, Schulz-Kuhnt A, Stahl A, Schulze LL, Ullrich K, Merz SF, Bornemann L, Gunzer M, Watson AJM, Neufert C, Atreya I, Neurath MF, Zundler S. Non-classical monocyte homing to the gut via alpha4beta7 integrin mediates macrophage-dependent intestinal wound healing. Gut. 2020 Feb;69(2):252-263. doi: 10.1136/gutjnl-2018-316772. Epub 2019 May 15. PMID 31092589
- [Background] Lee SH, Walshe M, Oh EH, Hwang SW, Park SH, Yang DH, Byeon JS, Myung SJ, Yang SK, Greener T, Weizman AV, Silverberg MS, Ye BD. Early Changes in Serum Albumin Predict Clinical and Endoscopic Outcomes in Patients With Ulcerative Colitis Starting Anti-TNF Treatment. Inflamm Bowel Dis. 2021 Aug 19;27(9):1452-1461. doi: 10.1093/ibd/izaa309. PMID 33269403
- [Background] Kim J, Yoon H, Kim N, Lee KM, Jung SA, Choi CH, Kim ES, Jung Y, Eun CS, Kim TO, Kang SB, Kim YS, Seo GS, Lee CK, Im JP, Park SJ, Park DI, Ye BD. Clinical Outcomes and Response Predictors of Vedolizumab Induction Treatment for Korean Patients With Inflammatory Bowel Diseases Who Failed Anti-TNF Therapy: A KASID Prospective Multicenter Cohort Study. Inflamm Bowel Dis. 2021 Nov 15;27(12):1931-1941. doi: 10.1093/ibd/izaa361. PMID 33501935
- [Background] Bandres-Ciga S, Saez-Atienzar S, Kim JJ, Makarious MB, Faghri F, Diez-Fairen M, Iwaki H, Leonard H, Botia J, Ryten M, Hernandez D, Gibbs JR, Ding J, Gan-Or Z, Noyce A, Pihlstrom L, Torkamani A, Soltis AR, Dalgard CL; American Genome Center; Scholz SW, Traynor BJ, Ehrlich D, Scherzer CR, Bookman M, Cookson M, Blauwendraat C, Nalls MA, Singleton AB; International Parkinson Disease Genomics Consortium. Large-scale pathway specific polygenic risk and transcriptomic community network analysis identifies novel functional pathways in Parkinson disease. Acta Neuropathol. 2020 Sep;140(3):341-358. doi: 10.1007/s00401-020-02181-3. Epub 2020 Jun 29. PMID 32601912
- [Background] Reay WR, Atkins JR, Carr VJ, Green MJ, Cairns MJ. Pharmacological enrichment of polygenic risk for precision medicine in complex disorders. Sci Rep. 2020 Jan 21;10(1):879. doi: 10.1038/s41598-020-57795-0. PMID 31964963